CLINICAL TRIAL: NCT01316484
Title: Protocol for the Patient Understanding (Cognitive Debriefing) of a Modified Gastroparesis Cardinal Symptom Index (GCSI) Daily Diary
Brief Title: Patient Understanding (Cognitive Debriefing) of a Daily Diary of Gastroparesis Symptoms
Status: Completed | Type: Observational
Sponsor: Tranzyme, Inc. (Industry)
Responsible Party: Robert P. Venuti, Director, Clinical Development, Tranzyme, Inc
Other Study IDs: TZP-QM-001
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Diabetes Mellitus; Gastroparesis
Keywords: Cognitive Debriefing
MeSH Terms: conditions — Diabetes Mellitus; Gastroparesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment: Adult subjects with diabetes mellitus and a diagnosis of gastroparesis

SUMMARY:
The primary objective of the study is to evaluate how patients with gastroparesis interpret the instructions, item content, and response options of a daily diary questionnaire designed to assess the key symptoms of gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has Type 1 or Type 2 diabetes mellitus
2. Subject is 18 to 70 years old
3. Subject has chronic, active symptoms of gastroparesis for at least the past three months
4. Subject has confirmed delayed gastric emptying by scintigraphy, a breath test, or the SmartPill® wireless motility capsule
5. Subject can speak and read English
6. Subject is able to give his/her informed consent

Exclusion Criteria:

1. Subject has a cognitive, psychological or other (e.g., visual) impairment that would interfere with completing the study visit

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital/Clinic Database
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Qualitative, Content Analysis of Cognitive Debriefing Data | 90-minute interview
  The cognitive debriefing data will be content analyzed for patient understanding of the concepts in the questionnaire and interpretation of the items' content.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Parkman, MD, Principal Investigator — Temple University Health Sciences Center; Tuba Esfandyari, MD, Principal Investigator — University of Kansas Medical Center; Irene Sarosiek, MD, Principal Investigator — Texas Tech University Health Sciences Center; Kenneth Koch, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Temple University Health Sciences Center, Philadelphia, Pennsylvania
  - Texas Tech University Health Sciences Center, El Paso, Texas